CLINICAL TRIAL: NCT07407205
Title: Tumor Mutational Burden, Liquid Biopsy, Angiogenic Factors and Magnetic Resonance Perfusion in Predicting Response to Chemoradiotherapy in HPV-Negative Oropharyngeal Squamous Cell Carcinoma and Disease Course After Treatment
Brief Title: Tumor Mutational Burden, Liquid Biopsy, Angiogenic Factors and DCE-MRI Perfusion in HPV-Negative Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OI-HPVNEG-OPC-TMB-2019; ARRS P3-0307 (Other: ARRS (Slovenian Research Agency))
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; HPV-Negative Oropharyngeal Cancer
Keywords: HPV-negative; oropharyngeal cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms | interventions — Chemoradiotherapy; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent Chemoradiotherapy (Experimental): Patients with HPV-negative oropharyngeal squamous cell carcinoma treated with standard concurrent chemoradiotherapy. Participants undergo additional diagnostic procedures including blood sampling for liquid biopsy biomarkers and dynamic contrast-enhanced MRI perfusion imaging for evaluation of predictive and prognostic markers.
  Interventions: Procedure: Concurrent Chemoradiotherapy; Diagnostic Test: Dynamic Contrast-Enhanced MRI Perfusion (DCE-MRI)

INTERVENTIONS:
Procedure: Concurrent Chemoradiotherapy — Standard-of-care concurrent chemoradiotherapy administered for HPV-negative oropharyngeal squamous cell carcinoma according to institutional treatment protocols.
Diagnostic Test: Dynamic Contrast-Enhanced MRI Perfusion (DCE-MRI) — Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) perfusion performed before and/or during treatment to obtain quantitative perfusion parameters and evaluate their predictive value for treatment response.

SUMMARY:
This prospective interventional study evaluates the predictive value of tumor mutational burden, liquid biopsy biomarkers (including circulating tumor DNA), angiogenic factors, and dynamic contrast-enhanced magnetic resonance (MR) perfusion imaging in patients with HPV-negative oropharyngeal squamous cell carcinoma treated with concurrent chemoradiotherapy. The aim is to improve prediction of treatment response and disease course after treatment, support decision-making regarding optimal therapy, and potentially reduce the number of imaging examinations required during follow-up.

DETAILED DESCRIPTION:
Patients with HPV-negative oropharyngeal squamous cell carcinoma treated with standard concurrent chemoradiotherapy are prospectively included in this study. The study investigates tumor mutational burden and specific somatic mutations in tumor tissue, as well as circulating tumor DNA (ctDNA) and other molecular biomarkers obtained through liquid biopsy. In addition, angiogenic factors in plasma and microRNA in extracellular vesicles are analyzed and compared with quantitative parameters obtained from dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) perfusion.

The main objective is to gain additional insight into tumor biology during and after chemoradiotherapy and to identify prognostic and predictive biomarkers associated with treatment response and disease progression. The study also aims to assess whether biomarker-based monitoring may reduce the need for repeated imaging examinations while maintaining accurate evaluation of treatment response and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Histologically confirmed HPV-negative oropharyngeal squamous cell carcinoma

Planned treatment with concurrent chemoradiotherapy

Ability to undergo MRI examination

Signed informed consent

Exclusion Criteria:

HPV-positive oropharyngeal carcinoma

Contraindications for MRI

Severe comorbidities preventing chemoradiotherapy

Pregnancy or breastfeeding

Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of Biomarkers and DCE-MRI for Response to Chemoradiotherapy | Up to 6 months after completion of concurrent chemoradiotherapy
Predictive Value of Biomarkers and DCE-MRI for Response to Chemoradiotherapy | Up to 6 months after completion of concurrent chemoradiotherapy
  Association of tumor mutational burden, somatic mutations (tumor tissue and/or ctDNA), liquid biopsy biomarkers (ctDNA, angiogenic factors, microRNA in extracellular vesicles), and dynamic contrast-enhanced MRI (DCE-MRI) perfusion parameters with treatment response after concurrent chemoradiotherapy in HPV-negative oropharyngeal squamous cell carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No